CLINICAL TRIAL: NCT03643016
Title: Improving EPilepsy Surgery Management and progNOsis Using Virtual Epileptic Patient Software (VEP)
Acronym: EPINOV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018-41
Record Dates: First submitted 2018-08-21; First posted 2018-08-22 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-09

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group with Virtual Epileptic Patient brain access data (Experimental)
  Interventions: Other: Surgical strategy based on a software
- Group without Virtual Epileptic Patient brain access data (No Intervention)

INTERVENTIONS:
Other: Surgical strategy based on a software — Surgical strategy décision based on a software
  Arms: Group with Virtual Epileptic Patient brain access data

SUMMARY:
Every year, thousands of patients worldwide with drug resistant focal epilepsy (DRE) undergo resective brain surgery with the aim of achieving seizure freedom.

Despite technical advances over the last 50 years, the success rate of epilepsy surgery in terms of seizure freedom has not greatly improved, remaining overall at around 50%. Depending on features of individual cases, presurgical evaluation includes a first phase of non-invasive data including video-EEG recordings, magnetoencephalography, structural and functional neuroimaging and neuropsychological evaluation. If these investigations do not allow adequate localization of likely region of seizure organization in the brain (the epileptogenic zone, EZ), then a second invasive phase using intracerebral EEG recording may be necessary (stereoelectroencephalography, SEEG). Interpretation of SEEG remains difficult in many cases, in particular since seizure onset is often characterized by discharges that very rapidly involve several distinct brain regions.

No reliable measuring instrument currently exists to combine the various prognostic factors for a given patient. This leads to great uncertainty on an individual scale in predicting the effects of surgery. The mapping of epileptic networks in patients with DRE is an innovative scientifically-validated and clinically-tested method to significantly improve accuracy of SEEG and presurgical interpretation and guide surgical strategies in patients with DRE. Therefore, the investigators developed the Virtual Epilepsy Patient software. Retrospective study already demonstrated the pertinence of this approach in improving the anatomical mapping of epileptogenic networks. Now, the investigators aim to prospectively demonstrate the role of VEP during presurgical evaluation of DRE patients

ELIGIBILITY:
Inclusion Criteria:

* Patient or pediatric patient suffering from drug-resistant focal epilepsy.
* Standardized presurgical evaluation including medical history, scalp video-EEG, 3T MRI (DTI and rsMRI), FDG-PET, Neuropsychological tests.
* Inpatient in one of the participating centers for recording seizure during long term SEEG-monitoring.

Exclusion Criteria:

* Epilepsy surgery performed without the requirement of SEEG or contra-indication to epilepsy surgery.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 356 (Estimated)
Dates: Start 2019-06-26 (Actual); Primary Completion 2024-12-23 (Estimated); Study Completion 2025-12-23 (Estimated)

PRIMARY OUTCOMES:
Clinical success, defined as seizure free patient without disabling side effect (clinical judgment) at 12-month follow-up | 12 months
  Number of seizure (Engel I)

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Garrido-Pradalié, Study Director — Assitance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No